CLINICAL TRIAL: NCT00919178
Title: Phase I Evaluation of the Safety and Immunogenicity of rDEN4delta30 Lot# 109A, a Live Attenuated DEN4 Vaccine, in Healthy Flavivirus-naïve Adult Volunteers.
Brief Title: Safety of and Immune Response to DEN4 Vaccine Component Candidate for Dengue Virus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CIR 256
Record Dates: First submitted 2009-06-11; First posted 2009-06-12 (Estimated); Last update posted 2013-01-03 (Estimated); Status verified 2012-12

CONDITIONS: Dengue Shock Syndrome; Dengue Hemorrhagic Fever
Keywords: Dengue virus; Vaccine; DEN4; Dengue
MeSH Terms: conditions — Severe Dengue; Dengue

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Participants will receive a single immunization for Dengue virus serotype 4 (DEN4)
  Interventions: Biological: DEN4 Vaccine Candidate
- 2 (Placebo Comparator): Participants will receive a single immunization in the form of placebo resembling vaccine for DEN 4
  Interventions: Biological: DEN4 Vaccine Placebo

INTERVENTIONS:
Biological: DEN4 Vaccine Candidate — DEN4 Vaccine Candidate
  Participants will receive a single immunization on Study Day 0. Vaccine will be delivered by subcutaneous injection in the upper arm, at a volume of 0.5 mL.
  Arms: 1
Biological: DEN4 Vaccine Placebo — DEN4 Vaccine Placebo
  Participants will receive a single immunization on Study Day 0. Placebo will be delivered by subcutaneous injection in the upper arm, at a volume of 0.5 mL.
  Arms: 2

SUMMARY:
Infection with dengue viruses is one of the leading causes of hospitalization and death in children in several tropical Asian counties. The World Health Organization (WHO) estimates that these viruses are responsible for more than 50 million cases of dengue fever (DF) and approximately 0.5 million cases of the more severe disease, dengue hemorrhagic fever/ shock syndrome (DHF/DSS) annually. Because dengue viruses are endemic in most tropical and subtropical regions, keeping more than 2 billion persons at risk for acquiring dengue, the WHO has made development of a dengue vaccine a top priority.

The purpose of this study is to evaluate the safety and effectiveness of a candidate DEN4 vaccine aimed at preventing infection with dengue virus serotype 4.

DETAILED DESCRIPTION:
Dengue viruses are endemic in most tropical and subtropical regions of the world with more than 2 billion persons at risk for acquiring dengue. There are four serotypes of dengue virus (DEN 1, DEN 2, DEN 3, and DEN 4) each capable of causing dengue illness ranging from mild, self-limited febrile illness to life-threatening disease. Because previous infection with one dengue serotype can increase the risk for DHF/DSS following infection with a different serotype, immunization would ideally provide immunity against all four dengue viral serotypes.

Several live, attenuated dengue vaccines have been tested in Phase I and/or Phase II clinical trials. Although some have appeared promising in early trials, none have been able to meet the requirements for a safe and effective vaccine. Meeting these requirements has been particularly difficult when testing vaccines containing all four serotypes. The vaccine candidate in this study is live-attenuated rDEN4delta30, which will target the DEN4 serotype, it is a potential component for a future tetravalent dengue vaccine.

This is a double-blind, random assignment, placebo-controlled study in healthy, adult volunteers. The purpose of this study is to evaluate the safety and effectiveness of a single dose of DEN4 vaccine. Some participants will be receiving placebo as a comparative measure, to better assess vaccine-associated versus non vaccine-associated adverse events.

To qualify for participation in the study, volunteers will undergo an eligibility screening which will include medical history, physical exam, hematology testing, liver and renal function testing, coagulation studies, human immunodeficiency virus (HIV) and hepatitis B and C screening, urinalysis, and screening for pervious flavivirus infection. Urine pregnancy testing will also be required for female volunteers.

Duration of individual participation in the study is approximately 26 weeks following vaccination on Study Day 0. Volunteers will be randomly assigned to receive either rDEN4delta30 or placebo; 50 participants will receive the vaccine, 20 will receive placebo. On the day of vaccination, all volunteers will be reassessed by study personnel to ensure continued eligibility, vital signs will be taken, and a physical exam will be performed. Female participants will also have a pregnancy test and review of acceptable pregnancy prevention methods. Eligible participants will receive a vaccination of Study Day 0, followed by a 30 minute post vaccination assessment for adverse events. After vaccination, volunteers will be evaluated in the clinic approximately every other day for the first 16 days if study.

During the course of study, volunteers will have blood drawn and clinical evaluations performed on Study Days 21, 28, 42, and 180 post-vaccination. All participants will be asked to record oral temperatures 3 times a day for the first 16 days post-vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide informed consent
* Good general health as determined by physical examination, laboratory screening, and review of medical history
* Available for the duration of the study, approximately 26 weeks postvaccination
* Willing to use acceptable forms of birth control. More information on this criterion can be found in the study protocol.

Exclusion Criteria:

* Currently breast-feeding, or pregnant
* Evidence of clinically significant neurologic, cardiac, pulmonary, hepatic, rheumatologic, autoimmune, or renal disease by history, physical examination, and/or laboratory studies
* Behavioral, cognitive, or psychiatric disease that in the opinion of the Investigator affects the ability of the volunteer to understand and cooperate with the requirements of the study protocol
* Screening laboratory values of Grade 1 or above for absolute neutrophil count(ANC), ALT, and serum creatinine, as defined in this protocol
* Any other condition that in the opinion of the Investigator would jeopardize the safety or rights of a volunteer participating in the trial or would render the volunteer unable to comply with the protocol
* Any significant alcohol or drug abuse in the past 12 months which has caused medical, occupational, or family problems, as indicated by volunteer history
* History of a severe allergic reaction or anaphylaxis
* Severe asthma (emergency room visit or hospitalization within the last 6 months)
* Positive HIV-1 serology by screening and confirmatory assays
* Positive for hepatitis C virus (HCV) by screening and confirmatory assays
* Positive for hepatitis B virus (HBV) by hepatitis B surface antigen (HBsAg) screening
* Any known immunodeficiency syndrome
* Use of anticoagulant medications
* Use of corticosteroids (excluding topical or nasal) or immunosuppressive drugs within 42 days prior to or following vaccination. Immunosuppressive dose of corticosteroids is defined as 10 mg or more prednisone equivalent per day for 14 or more days.
* Receipt of a live vaccine within 28 days or a killed vaccine within the 14 days prior to vaccination or anticipated receipt of any vaccine during the 42 days following vaccination
* History of a surgical splenectomy
* Receipt of blood products within the past 6 months, including transfusions or immunoglobulin or anticipated receipt of any blood products or immunoglobulin during the 42 days following vaccination
* History or serologic evidence of previous dengue virus infection or other flavivirus infection (e.g., yellow fever virus, St. Louis encephalitis, West Nile virus)
* Previous receipt of a flavivirus vaccine (licensed or experimental)
* Receipt of any investigational agent in the 42 days before or after vaccination
* Volunteer has definite plans to travel to a dengue endemic area during the study

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2009-07; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Immunogenicity of vaccine candidate, as assessed by neutralizing antibody titers to DEN4 | At Weeks 4 and 6 following vaccination
Safety of vaccine candidate, as assessed by the frequency of vaccine-related adverse events, graded by severity | Throughout study

SECONDARY OUTCOMES:
Frequency, quantity, and duration of viremia following vaccination | Throughout study
Number of vaccinees infected with vaccine virus | Throughout study
Infectivity rates, safety, and immunogenicity of a single dose of candidate vaccine compared with previous rates from a previous lot of similar vaccine | Throughout study
Durability of antibody response | At 26 Weeks following vaccination
Phenotype of peripheral blood mononuclear cells at primary infection with the rDEN4delta30 vaccine | Throughout study
Immunopathological mechanism of vaccine-associated rash in those volunteers who are willing to undergo skin biopsy | Throughout study
Cellular immune response to primary infection with the rDEN4delta30 vaccine | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Anna Durbin, MD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health; Beth Kirkpatrick, MD, Principal Investigator — University of Vermont Vaccine Testing Center
Locations (2):
- United States (2):
  - Center for Immunization Research, Johns Hopkins School of Public Health, Baltimore, Maryland
  - University of Vermont Vaccine Testing Center, Burlington, Vermont

REFERENCES:
- [Background] Swaminathan S, Khanna N. Dengue: recent advances in biology and current status of translational research. Curr Mol Med. 2009 Mar;9(2):152-73. doi: 10.2174/156652409787581592. PMID 19275624
- [Background] Tan GK, Alonso S. Pathogenesis and prevention of dengue virus infection: state-of-the-art. Curr Opin Infect Dis. 2009 Jun;22(3):302-8. doi: 10.1097/QCO.0b013e328329ae32. PMID 19262377
- [Background] Wiwanitkit V. Dengue vaccines: a new hope? Hum Vaccin. 2009 Aug;5(8):566-7. doi: 10.4161/hv.5.8.8481. Epub 2009 Aug 18. PMID 19337028